CLINICAL TRIAL: NCT07253584
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Safety and Efficacy of Recombinant Human Anti-PCSK9 Monoclonal Antibody Injection (SAL003) in Combination With Statin Therapy in Patients With Hypercholesterolemia and Mixed Dyslipidemia
Brief Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Safety and Efficacy of SAL003 in Combination With Statin Therapy in Patients With Hypercholesterolemia and Mixed Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL003A302
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Hyperlipidemias, Hypercholesterolemia, Mixed Dyslipidemia
Keywords: Low-density lipoprotein cholesterol; PCSK9; SAL003
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): SAL003 140 mg
  Interventions: Drug: SAL003 140 mg
- Reference Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAL003 140 mg — SAL003 140 mg
  Arms: Test Group
Drug: Placebo — Placebo
  Arms: Reference Group

SUMMARY:
A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Study to Evaluate the Safety and Efficacy of Recombinant Fully Human Anti-PCSK9 Monoclonal Antibody Injection (SAL003) in Combination with Statin Therapy in Patients with Hypercholesterolemia and Mixed Dyslipidemia.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of SAL003, a recombinant fully human anti-PCSK9 monoclonal antibody, in Chinese patients with hypercholesterolemia and mixed dyslipidemia at very high or high cardiovascular risk who have not achieved target LDL-C levels despite stable, moderate- to high-intensity statin therapy (with or without ezetimibe).

Approximately 720 participants will be randomized in a 2:1 ratio to receive either SAL003 140 mg or matching placebo, administered subcutaneously every 4 weeks for 24 weeks. Following the double-blind period, all participants will enter an open-label extension period and receive SAL003 140 mg Q4W for an additional 28 weeks, with a total study duration of 52 weeks.

The primary efficacy endpoint is the percent change from baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24. Key secondary endpoints include the absolute change in LDL-C, the proportion of subjects achieving LDL-C target levels, and changes in other lipid parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 75 years.
* On a stable, moderate- to high-intensity statin regimen (with or without ezetimibe) for at least 4 weeks prior to screening.
* Fasting LDL-C above target levels per 2023 Chinese guidelines:

With ASCVD history: ≥1.4 mmol/L (Extreme Risk) or ≥1.8 mmol/L (Very High Risk). Without ASCVD history: ≥2.6 mmol/L (Moderate/High Risk) or ≥3.4 mmol/L (Low Risk).

Fasting triglycerides (TG) ≤ 5.6 mmol/L at screening/randomization.

* Provide signed informed consent.

Exclusion Criteria:

* Homozygous Familial Hypercholesterolemia (HoFH).
* Uncontrolled hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg).
* Significant cardiovascular event (e.g., MI, unstable angina, stroke, PCI, CABG) within 3 months prior to screening.
* Heart failure (NYHA Class III or IV) or LVEF <40% within 3 months.
* Severe renal impairment (eGFR <30 mL/min/1.73m²).
* Active liver disease or significant hepatic impairment (ALT/AST >2.5x ULN or TBiL >2x ULN).
* Uncontrolled diabetes (HbA1c >8.0%) or type 1 diabetes.
* Use of other lipid-lowering therapies (e.g., fibrates, niacin) within 3 months or any PCSK9 inhibitor within 6 months prior to screening.
* Known hypersensitivity to any component of the investigational product or other antibody therapies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Percent change of LDL-C | at Week 24
  Percent change from baseline in LDL-C at Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Zuyi Yuan, M.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No